CLINICAL TRIAL: NCT01266070
Title: A Pilot Trial of TKI 258 (Dovitinib) in Von Hippel-Lindau Syndrome
Brief Title: TKI 258 in Von Hippel-Lindau Syndrome (VHL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial met toxicity stopping rule
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0650; NCI-2011-00305 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2015-12

CONDITIONS: Von Hippel-Lindau Syndrome
Keywords: VHL; Hemangioblastoma; Tumor of the central nervous system; TKI258
MeSH Terms: conditions — von Hippel-Lindau Disease; Hemangioblastoma; Central Nervous System Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dovitinib (Experimental): 500 mg/day on a 5 day on, 2 day off schedule
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — 500 mg (5 capsules) daily by mouth on Days 1-5, 8-12, 15-19, and 22-26 of each 28-day cycle (i.e. 5 days on, 2 days off schedule).
  Other Names: TKI258

SUMMARY:
The goal of this clinical research study is to learn if dovitinib can safely be given to patients who have VHL with a measurable hemangioblastoma (tumor of the central nervous system). The effects of this drug on the disease will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Dovitinib is designed to perform several anti-tumor functions, including cutting off the blood supply to tumors.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 5 dovitinib capsules by mouth each day on Days 1-5, 8-12, 15-19, and 22-26 of each 28-day cycle.

You should take the dovitinib capsules with about a cup (8 ounces) of water and at least 1 hour before breakfast or at least 2 hours following breakfast.

If you have any side effects from the drug, tell the study doctor right away. The study doctor may then lower the dose or keep the dose level the same.

If you miss a dose of dovitinib on Days 1-4 (or 8-11, 15-18, or 22-25), you should not make up the dose on the same day. You should continue taking the drug as scheduled the following day. If you miss a dose on Day 5 (or 12, 19, or 26), you should skip the dose, rest 2 days, and begin dosing again as scheduled on Day 8 (or 15, 22, or 1 of the next cycle). The study doctor will tell you about any additional steps that should be taken if you miss a dose.

Every 4 weeks on this study is called a study "cycle."

Study Visits:

On Day 1 of Cycle 1, you will have an ECG.

On Day 14 (+/- 3 days) of Cycles 1 and 2:

-Blood (about 3 teaspoons) will be drawn for routine tests. This blood testing may be done at your local doctor's office and faxed to MD Anderson. You will be provided instructions about how to fax laboratory test results.

On Day 1 of Cycles 3 and Beyond (+/- 3 days), blood (about 3 teaspoons) will be drawn for routine tests.

Every 8 weeks (+/- 3 days):

* Any changes to your medical history since your last visit will be recorded.
* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any drugs or treatments you may be receiving.
* Your performance status will be recorded.
* You will be asked about any side effects that you have had since your last visit.

At the End of Cycles 2 and 4:

* You will have CT scans and MRI scans to check the status of the disease.
* If the doctors know or suspect that VHL is affecting your eyes, you will have an eye exam.

Length of Study:

You may continue taking the study drugs for as long as you are benefiting. You will be taken off study if the disease gets worse or intolerable side effects occur.

Early Withdrawal /End of Treatment Visit:

* About 30 days after you stop taking study drug, you will have the following procedures:
* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects that you may have had since your last visit.
* Blood (about 3 teaspoons) will be drawn for routine tests.
* You will have CT scans and MRI scans to check the status of the disease.
* If the doctors know or suspect that VHL is affecting your eyes, you will have an eye exam.

About 24 weeks after your last dose of study drug, you will have the following procedures:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will have follow-up imaging scans to check the status of the disease.
* Blood (about 3 teaspoons) will be collected for routine tests.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects that you may have had since your last visit.

This is an investigational study. Dovitinib is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 25 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have genetically confirmed Von Hippel-Lindau (VHL) disease or patients with a clinical diagnosis of VHL.
2. At least one of the following measurable hemangioblastomas which is undergoing surveillance and the patient is not at immediate risk of needing intervention for this or other lesions. a.) Brain: asymptomatic hemangioblastoma, > 0.5 cm; b.) Spine: asymptomatic hemangioblastoma, > 0.5 cm; c.) Renal: solid mass suspicious for RCC >/=1 cm or cystic mass >/=1 cm; d.) Pancreas: solid mass >/=1cm and < 3 cm suspicious for neuroendocrine tumor; e.) Eye: asymptomatic peripapillary and/or macular hemangioblastoma, any size f. Adrenal: Pheochromocytoma greater than 1cm in size. NOTE: Biopsy is not required given the known natural history in the setting of a positive genetic test.
3. Allowable prior therapy: a.) Patients having undergone prior therapy for VHL lesions may enroll as long as other criteria are met. Previously radiated lesions may not be considered as target lesions unless they demonstrate unequivocal evidence of growth; b.) Major surgery, chemotherapy or radiation therapy completed > 4 weeks prior to starting the study treatment.
4. Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of dovitinib in patients < 18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable
5. ECOG performance status </= 2
6. Patients must have normal organ and marrow function as defined below: a.) Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) </=2.5 x local laboratory upper limit of normal (ULN) are due to underlying malignancy; b.) Total serum bilirubin </=1.5 x ULN; c.) Absolute neutrophil count (ANC) >/= 1500/mcL; d.) Platelets >/=100,000/mcL; e.) Hemoglobin >/= 9.0 g/dL; f.) Serum creatinine < 1.5 x ULN; g) WBC >/= 3,000/mcl
7. Males (that have not been sterilized) and females of childbearing potential (female that has not be amenorrheic for at least 1 year or that has not surgically sterilized) must agree to use double-barrier birth control or abstinence while on the protocol treatment
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to starting study treatment or those who have not recovered (</= Grade 1 )from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents.
3. Patients with any metastatic disease of any kind.
4. NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment.
5. Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
6. Ongoing cardiac dysrhythmias of NCI CTCAE grade >/= 2.
7. Prolonged QTc interval on baseline EKG > 470ms.
8. Hypertension that cannot be controlled by medications (>140/90 mm Hg despite optimal medical therapy).
9. LVEF assessed by 2-D echocardiogram (ECHO) < 50% or lower limit of normal (whichever is higher) or multiple gated acquisition scan ( MUGA) < 45% or lower limit of normal (whichever is higher).
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Pregnant women are excluded from this study because dovitinib has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dovitinib, breastfeeding should be discontinued if the mother is treated with dovitinib.
12. Known HIV-positive patients taking combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dovitinib. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
13. Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception. Highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 8 weeks after the end of study treatment. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test </= 14 days prior to starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Larcher A, Rowe I, Belladelli F, Fallara G, Raggi D, Necchi A, Montorsi F, Capitanio U, Salonia A; OSR VHL Program. Von Hippel-Lindau disease-associated renal cell carcinoma: a call to action. Curr Opin Urol. 2022 Jan 1;32(1):31-39. doi: 10.1097/MOU.0000000000000950. PMID 34783716
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 16, 2012 to January 30, 2014. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Dovitinib: Dovitinib oral 500 mg/day on a 5 day on, 2 day off schedule (Days 1-5, 8-12, 15-19, and 22-26) of each 28-day cycle
Period: Overall Study
Arm/Group | Dovitinib
Started | 6
Completed | 2
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dovitinib
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 44 [18 to 62]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Most Frequent & Most Serious Adverse Events: Safety of Dovitinib for 6 Months
Description: Most frequent & Most Serious Adverse Events: Safety of treatment with Dovitinib for 6 months in participants with VHL who have a measurable hemangioblastoma undergoing surveillance evaluated by toxicity scored using Common Toxicity Criteria (CTC) Version 4.0.
Time Frame: Every 2 cycles (approximately 8 weeks) for 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 6
Participants
  Alanine aminotransferase increased | 6
  Alkaline phosphatase increased | 6
  Aspartate aminotransferase increased | 6
  Diarrhea | 5
  Dyspepsia | 3
  GGT Increased | 5
  Hyperglycemia | 4
  Hyperkalemia | 4
  Mucositis oral | 4
  Nausea | 6
  Rash maculo-papular | 6
  White Blood cell decreased | 5

2. Secondary Outcome: Number of VHL Participants With Response at 6 Months
Description: Efficacy of treatment with dovitinib for 6 months in patients with VHL who have a measurable lesion evaluated by response using RECIST (Response Evaluation Criteria in Solid Tumors): Complete Response, Partial Response, Progressive Disease or Stable Disease.
Time Frame: Every 2 cycles (approximately 8 weeks) for 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected through 28 day treatment cycle, up to 6 months.
Arm/Group | Dovitinib
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=6)
Abdominal pain (General disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (12)
Alkaline phosphatase increased (Investigations) | 6 (7)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Blurred vision (Eye disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 2 (2)
GGT increased (Investigations) | 5 (5)
Headache (Nervous system disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Lipase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (9)
Neutrophil count decreased (Investigations) | 2 (2)
Pain (Dorsum of Left Foot) (General disorders) | 1 (1)
Pain (Tooth Pain) (General disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (13)
Serum amylase increased (Investigations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes